CLINICAL TRIAL: NCT02973022
Title: A Community Based Approach to Reducing Rural Cancer Disparities, Aim 2
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: UW16048; 2016-0941 (Other: Institutional Review Board); A534253 (Other: UW Madison); SMPH\MEDICINE\GEN INT MD (Other: UW Madison); NCI-2019-06442 (Registry Identifier: NCI Trial ID); NCT02886325 (obsolete NCT alias)
Record Dates: First submitted 2016-11-21; First posted 2016-11-25 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Community CC&S Group: Once participants are randomized, they will be given survey 1. The intervention group in the community will be exposed to the modified CC&S educational sessions in a series of 2 one hour and 15 minute sessions on consecutive Monday nights. A free meal will be provided at both educational sessions. Childcare will be provided for community sessions. Once the final educational session is completed, all participants will be given survey 2.
  Interventions: Other: CC&S
- Community Control Group: Once participants are randomized, they will be given survey 1. The control group in the community will be exposed to a nutrition education program in a series of 2 one hour and 15 minute sessions on consecutive Monday nights. A free meal will be provided at both educational session. Childcare will be provided for community sessions. Once the final educational session is completed, all participants will be given survey 2.
- ACEC CC&S Group: Once participants are randomized, they will be given survey 1. The intervention group at ACEC (Adams-Columbia Electric Company) will be exposed to the modified CC&S educational sessions in a series of 6 thirty minute sessions before the work day begins over the course of several weeks. The researchers anticipate that two sessions will occur per week and therefore the delivery of the whole intervention will take 3 weeks. A free meal will be provided at all 6 educational sessions. Once the final educational session is completed, all participants will be given survey 2.
  Interventions: Other: CC&S
- ACEC Control Group: Once participants are randomized, they will be given survey 1. The control group at ACEC will be exposed to a nutrition education program in a series of 6 thirty minute sessions before the work day begins over the course of several weeks. We anticipate that two sessions will occur per week and therefore the delivery of the whole intervention will take 3 weeks. A free meal will be provided at all 6 educational sessions. Once the final educational session is completed, all participants will be given survey 2.

INTERVENTIONS:
Other: CC&S — Three educational modules -- Cancer Basics, Cancer Prevention, and Cancer Screening -- intended to increase cancer awareness. The full CC&S curriculum is currently available at http://chdi.wisc.edu/cancer-clear-simple-curriculum-rural-adaptation.
  Other Names: Cancer Clear & Simple
  Groups: ACEC CC&S Group; Community CC&S Group

SUMMARY:
The aim of this study is to evaluate the impact of participation in Cancer Clear and Simple (CC&S) educational sessions on cancer prevention and screening. The researchers will recruit 60 community members: 30 will receive CC&S training (intervention group) and 30 will not (control group). All 60 will be surveyed about their intent to change their behavior at the beginning of the study and their actual behavior changes and their screening behavior 6 months after enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Wisconsin resident

Exclusion Criteria:

* None

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty ACEC employees and 30 residents of a rural Wisconsin county. The researchers will work to make sure the sample is representative of the community in regards to age, gender, and employments status.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Change in behavioral intent | Up to 3 weeks
  All 60 participants (30 intervention, 30 control group) will be surveyed about their intent to change their behavior at the beginning of the study and their actual behavior changes and their cancer screening behavior 6 months after enrollment in the study.

SECONDARY OUTCOMES:
Change in cancer knowledge | Up to 6 months
  Change in cancer knowledge measured before the educational session to after the session and duration of that knowledge as measured from right after the session to six months later.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jacobs, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252